CLINICAL TRIAL: NCT06516237
Title: Relationships Between Intestinal Ultrasound Parameters and Elastography Measurements With Histopathologic Findings in a Prospective Cohort of Patients With Ulcerative Colitis: Development of Novel Imaging and Molecular Biomarkers of Fibrosis
Brief Title: Development of Novel Imaging and Molecular Biomarkers of Fibrosis in Patient With Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Mariangela Allocca, Gastroenterologist, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Strictur-US
Record Dates: First submitted 2024-06-10; First posted 2024-07-23 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: 50 Consecutive adult (18 years of age and older) patients with an established diagnosis (> 3 months) of ulcerative colitis irrespective to state of disease and treatment, undergoing routine investigations by colonoscopy or sigmoidoscopy(according to the current standard of care indications and ECCO guidelines), will be enrolled and undergone routine biopsies in the distal colon and intestinal ultrasound with Shear wave elastography measurements. In addition, up to 8 biopsies will be performed, at clinical judgment, in distal colon to determine molecular and epigenetic biomarkers. Any medication will be kept stable in the interval between the two procedures.
Masking Description: Ultrasound and endoscopy will be performed within 7 days in blinded fashion, where the ultrasound operators will be blinded to clinical and endoscopic findings and the endoscopist will be blinded of the clinical and ultrasound findings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- to develop novel imaging and molecular biomarkers of fibrosis (Other): 50 Consecutive adult (18 years of age and older) patients, undergoing routine investigations by colonoscopy or sigmoidoscopy, will be enrolled and undergone routine biopsies in the distal colon and intestinal ultrasound with Shear wave elastography measurements.
  Interventions: Procedure: to determine molecular and epigenetic biomarkers

INTERVENTIONS:
Procedure: to determine molecular and epigenetic biomarkers — In addition, up to 8 biopsies will be performed, at clinical judgment, in distal colon to determine molecular and epigenetic biomarkers.

SUMMARY:
Prospective multicenter interventional non-randomized cross-sectional study. Ultrasound operators will be blinded to clinical and endoscopic findings and the endoscopist will be blinded of the clinical and ultrasound findings.

This study aims to develop novel imaging and molecular biomarkers of fibrosis, through the use of intestinal ultrasound and shear wave elastography, using histologic specimens obtained by endoscopic biopsies as reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Adult, 18 years of age and older,
* Established diagnosis (> three months) of ulcerative colitis,
* Performing colonoscopy, according to current standards of care and ECCO guidelines,
* Ability to understand and comply with the study procedure and sign an informed consent form

Exclusion Criteria:

* Pregnancy,
* presence of ascites, active infections, any contraindication to colonoscopy (e.g. intolerance to preparation, severe flare),
* inability to undergo intestinal ultrasound within the time set by the study,
* poor quality of ultrasound imaging (due to luminal gas or body habitus), or a diagnosis of malignancy in the pathological specimen.
* subjects who needs to change therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
To correlate ultrasound findings with histopathological elements of lesions | 1 day
  To correlate ultrasound findings with histopathological elements of lesions obtained by biopsies of the distal colon during routine investigations by colonoscopy or sigmoidoscopy, as the reference standard: specifically, Hematoxylin and Eosin (H&E) staining for inflammation, Immunostaining of alfa-smooth muscle actin (aSMA) for muscular hypertrophy, and Sirius red special staining for collagen deposition

SECONDARY OUTCOMES:
To correlate shear wave elastography measurements with histopathological elements of lesions | 1 day
  To correlate shear wave elastography measurements with histopathological elements of lesions, Hematoxylin and Eosin (H&E) staining for inflammation, Immunostaining of alfa-smooth muscle actin (aSMA) for muscular hypertrophy, and Sirius red special staining for collagen deposition

OTHER OUTCOMES:
To correlate ultrasound findings and shear wave elastography measurements with molecular and epigenetic characteristics at single cell resolution | 1 day
  To correlate ultrasound findings and shear wave elastography measurements with molecular and epigenetic characteristics at single cell resolution

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milano, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No